CLINICAL TRIAL: NCT00477737
Title: Early Cardioprotective Effect of Sevoflurane on Left Ventricular Performance During Coronary Artery Bypass Grafting on a Beating Heart
Brief Title: Early Cardioprotective Effect of Sevoflurane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARPRO10
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Artery Disease; Off Pump Coronary Artery Bypass Surgery
Keywords: cardioprotection; sevoflurane; esophageal Doppler; thermodilution; coronary artery bypass
MeSH Terms: conditions — Coronary Artery Disease | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sevoflurane
Drug: propofol

SUMMARY:
In vitro studies and in vivo animal experiments have shown that halogenated volatile anesthetics have a protective effect on the ischemic myocardium. In clinical settings however, anesthetic preconditioning may be of more interest. The aim of our study was to evaluate the cardioprotective effect of sevoflurane in patients undergoing off-pump coronary artery bypass surgery. We proposed that a cardioprotective effect of sevoflurane would save myocardial function, which we measured acceleration by esophageal Doppler and cardiac index with bolus thermodilution methods, both during brief ischemia and reperfusion.

DETAILED DESCRIPTION:
Studies have been performed on human patients undergoing CABG surgery with cardiopulmonary bypass (CPB). Only a few studies however have evaluated the effects of volatile anesthetics during coronary artery bypass grafting on a beating heart (OPCABG) with conflicting results as far as cardiac biomarker release is concerned.

Because CPB is known to have a profound impact on cardiac function, studies performed on patients scheduled for OPCABG could evaluate more specifically the effects of the anesthetic agents themselves. Patients undergoing OPCABG have a predictable and predefined ischemic zone during surgery and represent an extremely interesting and safe model for the study of ischemia and cardiac damage in humans.

Presently, there is still no consensus on the method of administration of volatile anesthetics, including the time to begin administration, its duration, the dosage and selection of volatile anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* the degree I or II of Cardiac Anesthesia Risk Evaluation score
* angiographically verified coronary artery disease
* left ventricular ejection fraction higher than 40%

Exclusion Criteria:

* atrioventricular conduction disturbances
* previously ventricular arrhythmias requiring antiarrhythmic treatment
* atrial fibrillation with rapid ventricular response
* myocardial infarction or stroke within 6 months
* diabetes mellitus
* end-stage of obstructive or restrictive pulmonary disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate cardiac function with measuring of hemodynamic parameters | Measurements were performed at the following intervals: 5 minutes after anesthesia induction; at the beginning of ischemia; 15 minutes after ischemia; 15 minutes after sternum closure

CONTACTS AND LOCATIONS:
Overall Officials: Ino Husedzinovic, MD PhD Prof, Principal Investigator — Anesthesiology and Intensive Medicine
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Derived] Huseidzinovic I, Barisin S, Bradic N, Milanovic R. Early cardioprotective effect of sevoflurane on left ventricular performance during coronary artery bypass grafting on a beating heart: randomized controlled study. Croat Med J. 2007 Jun;48(3):333-40. PMID 17589976